CLINICAL TRIAL: NCT01082848
Title: Efficacy of Aripiprazole in the Treatment of Anorexia Nervosa in Teenagers: a Pilot, Randomised, Double Blind, Placebo-controlled Clinical Trial
Brief Title: ARIpiprazole in Anorexia NErvosa
Acronym: ARIANE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, Dr, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARIANE; 2009-010082-23 (EudraCT Number)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aripiprazole (Experimental)
  Interventions: Drug: aripiprazole
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aripiprazole — 10 mg QD during 26 weeks
  Arms: aripiprazole
Drug: placebo — QD during 26 weeks
  Arms: placebo

SUMMARY:
Evidence is lacking on the effects of different psychotropic drugs in the treatment of anorexia nervosa (AR). However, HVA levels seem to be elevated in this disease, therefore suggesting a role for drugs with a partial agonist profile on dopaminergic receptors. This is a pilot study assessing the effects of aripiprazole in teenagers with AR, compared with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* age between 12 and 18
* diagnostic criteria for anorexia Nervosa (DSM-IV-TR (includes BMI below 17.5kg/m2 and above 14 kg/m2) confirmed by a Psychiatrist and validated by K-SADS-PL interview
* severity criteria requiring Hospital admission
* Consent given by parents and patients

Exclusion Criteria:

* psychotic illness
* antipsychotic therapy at inclusion
* pregnancy and breastfeeding
* antipsychotic drug allergy
* prior head trauma, malignant neuroleptic syndrome or epilepsy
* relevant comorbidities requiring therapy
* detection of abuse drugs in urine test
* treatment with neuroleptic, antidepressant or mood stabilizers during 2 weeks prior to randomization (4 weeks in case of fluoxetine)
* suicidal or homicidal thoughts
* IQ below 70

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Inventory-2 | 6 months
Eating attitudes test (EAT) | 6 months
Brown Assessment of Beliefs Scale (BABS) | 6 months

SECONDARY OUTCOMES:
BMI | 6 months
  Body mass index
BDI | 6 months
  Beck Depression Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Catalonia, Spain